CLINICAL TRIAL: NCT04835714
Title: A Phase I Open-label Dose Escalation Trial of BI 1701963 as Monotherapy and in Combination With BI 3011441 in Patients With KRAS Mutated Advanced or Metastatic Solid Tumours
Brief Title: A Study to Find a Safe and Effective Dose of BI 1701963 Alone and in Combination With BI 3011441 in Patients With Advanced Cancer and a Certain Mutation (Kirsten Rat Sarcoma Viral Oncogene Homologue [KRAS])
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 1432-0006
Record Dates: First submitted 2021-04-06; First posted 2021-04-08 (Actual); Last update posted 2023-02-01 (Actual); Status verified 2023-01

CONDITIONS: Solid Tumors, KRAS Mutation

STUDY DESIGN:
Masking Description: Description to randomisation:
  In Part A and Part B no randomisation will be performed. In Part C and Part D randomisation will be performed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Part A with Monotherapy dose escalation (Experimental)
  Interventions: Drug: BI 1701963
- Part B with Combination therapy dose escalation (Experimental)
  Interventions: Drug: BI 1701963; Drug: BI 3011441
- Part C with Combination therapy dose confirmation (Experimental)
  Interventions: Drug: BI 1701963; Drug: BI 3011441
- Part D with Combination therapy dose expansion (Experimental)
  Interventions: Drug: BI 1701963; Drug: BI 3011441

INTERVENTIONS:
Drug: BI 1701963 — BI 1701963
Drug: BI 3011441 — BI 3011441
  Arms: Part B with Combination therapy dose escalation; Part C with Combination therapy dose confirmation; Part D with Combination therapy dose expansion

SUMMARY:
This is a study in adults with advanced cancer (solid tumours including non-small cell lung cancer and colorectal cancer) in whom previous chemotherapy was not successful. People who have a tumour with a KRAS mutation can participate in the study. A KRAS mutation makes cancer grow faster.

The study tests 2 medicines called BI 1701963 and BI 3011441. BI 1701963 and BI 3011441 prevent activation of KRAS.

The purpose of this study is to find out the highest dose of BI 1701963 alone and in combination with BI 3011441 the participants can tolerate. Another purpose is to check whether BI 1701963 in combination with BI 3011441 is able to make tumours shrink.

Participants can stay in the study as long as they benefit from treatment and can tolerate it. During this time, they get tablets of BI 1701963 and capsules of BI 3011441 once daily. The doctors regularly monitor the size of the tumour. Doctors also regularly record any unwanted effects and check participants' health.

ELIGIBILITY:
Inclusion Criteria:

* Previously-identified activating Kirsten rat sarcoma viral oncogene homologue (KRAS) mutation in tumour tissue or blood prior to screening. Activating mutations may include but are not limited to: KRAS mutations in expressed region (exon) 2 (G12, G13), exon 3 (A59, Q61) and exon 4 (K117, A146).
* Provision of archival tumour tissue, if available, to confirm retrospectively KRAS mutation status and for biomarker assessment
* At least one target lesion that can be measured per Response Evaluation Criteria In Solid Tumours (RECIST) version 1.1. In patients who only have one target lesion, and a biopsy of the lesion is required, the baseline imaging must be performed at the earliest two weeks after the biopsy.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 at screening
* Adequate organ function at screening as follows:

  * Absolute neutrophil count (ANC) ≥1.5 x 109/L; hemoglobin ≥9.0 g/dL; platelets ≥100 x 109/L without the use of haematopoietic growth factors or recent transfusion
  * Total bilirubin ≤1.5 times the upper limit of normal (ULN), or ≤4 x ULN for patients who are known to have Gilbert's syndrome.
  * Creatinine ≤1.5 x ULN. If creatinine is >1.5 x ULN, patient is eligible if concurrent glomerular filtration rate (GFR) ≥50 mL/min (measured or calculated by Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) formula).
  * Aspartate transaminase (AST) and alanine transaminase (ALT) ≤3 x ULN if no demonstrable liver metastases, or ≤ 5 x ULN if transaminase elevation is attributable to liver metastases.
* Age ≥18 years of age, or over the legal age of consent as required by local legislation at informed consent.
* Recovery from any previous therapy related toxicity to Common Terminology Criteria for Adverse Events (CTCAE) Grade ≤1 at Cycle 1 Day 1 (except for alopecia, stable sensory neuropathy must be CTCAE Grade ≤2 and except for amenorrhea/menstruation related disorders of any grade) before the first dose.
* Signed and dated written informed consent in accordance with Good Clinical Practice (GCP) and local legislation prior to admission to the trial.

Further inclusion criteria apply.

Exclusion Criteria:

* Previous anticancer chemotherapy or anticancer immunotherapy within 3 weeks of the first administration of trial drug. Previous anticancer hormonal treatment within 2 weeks of the first administration of trial drugs.
* Previous treatment with Rat sarcoma (RAS), Mitogen-activated protein kinase (MAPK) or Son of Sevenless 1 (SOS1) targeting agents
* Radiotherapy within 4 weeks prior to start of treatment except as follows

  * Palliative radiotherapy to regions other than the chest is allowed up to 2 weeks prior to start of treatment
  * Single dose palliative radiotherapy for symptomatic metastasis within 2 weeks prior to start of treatment may be allowed but must be discussed with the sponsor.
* Major surgery (major according to the investigator's assessment) performed within 4 weeks prior to start of treatment or planned during the projected course of the trial, e.g. hip replacement.
* Previous treatment with any investigational agent(s) or targeted treatment within 28 days prior to start of treatment.
* Known history of hypersensitivity to any of the excipients of BI 1701963 tablets
* History or presence of cardiovascular abnormalities such as uncontrolled hypertension, congestive heart failure New-York-Heart-Assocation (NYHA) classification of ≥3, unstable angina or poorly controlled arrhythmia which are considered clinically relevant by the investigator; myocardial infarction within 6 months prior to start of treatment. Uncontrolled hypertension is defined as: Blood pressure (BP) measured in a rested and relaxed condition, where systolic BP ≥140 mmHg, or diastolic BP ≥90 mmHg, with or without medication.
* Left ventricular ejection fraction (LVEF) <50 %. Further exclusion criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2021-04-20 (Actual); Primary Completion 2022-01-18 (Actual); Study Completion 2022-01-18 (Actual)

PRIMARY OUTCOMES:
Number of patients with dose-limiting toxicities (DLTs) in the Maximum tolerated dose (MTD) evaluation period in monotherapy (Part A) | Up to 28 days
Number of patients with dose-limiting toxicities (DLTs) in the Maximum tolerated dose (MTD) evaluation period in combination therapy (Part B) | Up to 28 days
Objective response (OR) defined as best overall response of confirmed complete response (CR) or confirmed partial response (PR) in combination therapy dose confirmation (Part C) | Up to 12 months
  Best overall response is defined according to Response Evaluation Criteria In Solid Tumours (RECIST) version 1.1 as assessed by the investigator and will consider all tumour assessments from first administration until disease progression or death (whichever occurs first) or last evaluable tumour assessment before start of subsequent anticancer therapy, loss to follow-up or withdrawal of consent.
Objective response (OR) defined as best overall response of confirmed complete response (CR) or confirmed partial response (PR) in combination therapy dose expansion (Part D) | Up to 12 months
  Best overall response is defined according to Response Evaluation Criteria In Solid Tumours (RECIST) version 1.1 as assessed by the investigator and will consider all tumour assessments from first administration until disease progression or death (whichever occurs first) or last evaluable tumour assessment before start of subsequent anticancer therapy, loss to follow-up or withdrawal of consent.

SECONDARY OUTCOMES:
Maximum plasma concentration (Cmax) of BI 1701963 after the first dose in monotherapy (Part A) | Up to 24 hours
Maximum plasma concentration (Cmax) of BI 1701963 after the first dose in combination therapy (Part B) | Up to 24 hours
Area under the plasma concentration-time curve over the time interval from 0 to the last quantifiable data point (AUC0-tz) of BI 1701963 after the first dose in monotherapy (Part A) | Up to 24 hours
Area under the plasma concentration-time curve over the time interval from 0 to the last quantifiable data point (AUC0-tz) of BI 1701963 after the first dose in combination therapy (Part B) | Up to 24 hours
Maximum plasma concentration at steady state (Cmax,ss) of BI 1701963 after multiple doses in monotherapy (Part A) | Up to 12 weeks
Maximum plasma concentration at steady state (Cmax,ss) of BI 1701963 after multiple doses in combination therapy (Part B) | Up to 12 weeks
Area under the concentration-time curve at steady state over the uniform dosing interval τ (AUCτ,ss) of BI 1701963 after multiple doses in monotherapy (Part A) | Up to 12 weeks
Area under the concentration-time curve at steady state over the uniform dosing interval τ (AUCτ,ss) of BI 1701963 after multiple doses in combination therapy (Part B) | Up to 12 weeks
Maximum plasma concentration (Cmax) of BI 3011441 after the first dose (Part B only) | Up to 24 hours
Area under the plasma concentration-time curve over the time interval from 0 to the last quantifiable data point (AUC0-tz) of BI 3011441 after the first dose (Part B only) | Up to 24 hours
Maximum plasma concentration at steady state (Cmax,ss) of BI 3011441 after multiple doses (Part B only) | Up to 12 weeks
Area under the concentration-time curve at steady state over the uniform dosing interval τ (AUCτ,ss) of BI 3011441 after multiple doses (Part B only) | Up to 12 weeks
Number of patients with Common Terminology Criteria for Adverse Events (CTCAE) Grade ≥3 treatment-related adverse events observed during the on-treatment period in combination therapy dose confirmation (Part C) | Up to 12 months
Number of patients with Common Terminology Criteria for Adverse Events (CTCAE) Grade ≥3 treatment-related adverse events observed during the on-treatment period in combination therapy dose expansion (Part D) | Up to 12 months
Maximum plasma concentration (Cmax) of BI 1701963 after the first dose in combination therapy dose confirmation (Part C) | Up to 24 hours
Maximum plasma concentration (Cmax) of BI 1701963 after the first dose in combination therapy dose expansion (Part D) | Up to 24 hours
Area under the plasma concentration-time curve over the time interval from 0 to the last quantifiable data point (AUC0-tz) of BI 1701963 after the first dose in combination therapy dose confirmation (Part C) | Up to 24 hours
Area under the plasma concentration-time curve over the time interval from 0 to the last quantifiable data point (AUC0-tz) of BI 1701963 after the first dose in combination therapy dose expansion (Part D) | Up to 24 hours
Maximum plasma concentration at steady state (Cmax,ss) of BI 1701963 after multiple doses in combination therapy dose confirmation (Part C) | Up to 12 weeks
Maximum plasma concentration at steady state (Cmax,ss) of BI 1701963 after multiple doses in combination therapy dose expansion (Part D) | Up to 12 weeks
Area under the concentration-time curve at steady state over the uniform dosing interval τ (AUCτ,ss) of BI 1701963 after multiple doses in combination therapy dose confirmation (Part C) | Up to 12 weeks
Area under the concentration-time curve at steady state over the uniform dosing interval τ (AUCτ,ss) of BI 1701963 after multiple doses in combination therapy dose expansion (Part D) | Up to 12 weeks
Maximum plasma concentration (Cmax) of BI 3011441 after the first dose in combination therapy dose confirmation (Part C) | Up to 24 hours
Maximum plasma concentration (Cmax) of BI 3011441 after the first dose in combination therapy dose expansion (Part D) | Up to 24 hours
Area under the plasma concentration-time curve over the time interval from 0 to the last quantifiable data point (AUC0-tz) of BI 3011441 after the first dose in combination therapy dose confirmation (Part C) | Up to 24 hours
Area under the plasma concentration-time curve over the time interval from 0 to the last quantifiable data point (AUC0-tz) of BI 3011441 after the first dose in combination therapy dose expansion (Part D) | Up to 24 hours
Maximum plasma concentration at steady state (Cmax,ss) of BI 3011441 after multiple doses in combination therapy dose confirmation (Part C) | Up to 12 weeks
Maximum plasma concentration at steady state (Cmax,ss) of BI 3011441 after multiple doses in combination therapy dose expansion (Part D) | Up to 12 weeks
Area under the concentration-time curve at steady state over the uniform dosing interval τ (AUCτ,ss) of BI 3011441 after multiple doses in combination therapy dose confirmation (Part C) | Up to 12 weeks
Area under the concentration-time curve at steady state over the uniform dosing interval τ (AUCτ,ss) of BI 3011441 after multiple doses in combination therapy dose expansion (Part D) | Up to 12 weeks
Duration of Objective Response (OR) in combination therapy dose confirmation (Part C) | Up to 12 months
  Duration of OR is defined as the time from first documented CR or PR until disease progression or death (whichever occurs first) among patients with OR.
Duration of Objective Response (OR) in combination therapy dose expansion (Part D) | Up to 12 months
  Duration of OR is defined as the time from first documented CR or PR until disease progression or death (whichever occurs first) among patients with OR.
Tumour shrinkage (in millimetres) in combination therapy dose confirmation (Part C) | Up to 12 months
  Tumour shrinkage (in millimetres) is defined as the difference between the minimum post-baseline sum of diameters of target lesions (longest for non-nodal lesions, short axis for nodal lesions) and the baseline sum of longest diameters of the same set of target lesions.
Tumour shrinkage (in millimetres) in combination therapy dose expansion (Part D) | Up to 12 months
  Tumour shrinkage (in millimetres) is defined as the difference between the minimum post-baseline sum of diameters of target lesions (longest for non-nodal lesions, short axis for nodal lesions) and the baseline sum of longest diameters of the same set of target lesions.
Progression-free survival (PFS) rate at 6 months in combination therapy dose confirmation (Part C) | Up to 6 months
  Based on PFS defined as the time from first administration until tumour progression according to RECIST 1.1 or death from any cause, whichever occurs earlier
Progression-free survival (PFS) rate at 6 months in combination therapy dose expansion (Part D) | Up to 6 months
  Based on PFS defined as the time from first administration until tumour progression according to RECIST 1.1 or death from any cause, whichever occurs earlier

CONTACTS AND LOCATIONS:
Locations (4):
- Japan (4):
  - Aichi Cancer Center Hospital, Aichi, Nagoya
  - National Cancer Center Hospital East, Chiba, Kashiwa
  - National Cancer Center Hospital, Tokyo, Chuo-ku
  - Japanese Foundation for Cancer Research, Tokyo, Koto-ku

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents, except for the following exclusions:
  1. studies in products where Boehringer Ingelheim is not the license holder;
  2. studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials;
  3. studies conducted in a single center or targeting rare diseases (because of limitations with anonymization).
  For more details refer to: https://www.mystudywindow.com/msw/datasharing

REFERENCES:
- See also: Related Info — https://www.mystudywindow.com/